CLINICAL TRIAL: NCT00465738
Title: Prospective, Randomized, Observer-blind, Parallel-group, Multi-center Trial to Assess Efficacy and Safety of Two Different Dilutions of incobotulinumtoxinA (Xeomin) in Patients With Upper Limb Spasticity
Brief Title: IncobotulinumtoxinA (Xeomin) for Upper Limb Spasticity
Acronym: NT-Spin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Central Medical Affairs, Merz Pharmaceuticals GmbH
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRZ 60201 - 0607 / 1
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Results first posted 2010-12-06 (Estimated); Last update posted 2010-12-31 (Estimated); Status verified 2010-12

CONDITIONS: Upper Limb Spasticity
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL (Experimental): incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kD), free from complexing proteins")(active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection; Mode of administration: intramuscular injection; The content of the vial was dissolved in 5.0 mL of sterile sodium chloride [NaCl] 0.9% solution without preservatives. Dilution with 5.0 mL resulted in a dose of 20 units per 1.0 mL.
  Interventions: Drug: incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kD), free from complexing proteins")
- incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL (Active Comparator): incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kD), free from complexing proteins")(active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection; Mode of administration: intramuscular injection; The content of the vial was dissolved in 2.0 mL sterile of NaCl 0.9% solution without preservatives. Dilution with 2.0 mL resulted in a dose of 50 units per 1.0 mL.
  Interventions: Drug: incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kD), free from complexing proteins")

INTERVENTIONS:
Drug: incobotulinumtoxinA (Xeomin, also known as "NT 201" or "Botulinum toxin type A (150 kD), free from complexing proteins") — active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins; powder for solution for injection; Mode of administration: intramuscular injection; The content of the vial was dissolved in 2.0 or 5.0 mL of sterile sodium chloride [NaCl] 0.9% solution without preservatives. Dilution with 2.0 or 5.0 mL resulted in a dose of 50 or 20 units per 1.0 mL.
  Other Names: incobotulinumtoxinA; Xeomin; NT 201; Botulinum toxin type A (150 kD), free from complexing proteins

SUMMARY:
This study will investigate the efficacy and safety of incobotulinumtoxinA (Xeomin) in the treatment of arm tightness (upper limb spasticity) using two different dilutions of incobotulinumtoxinA (Xeomin).

DETAILED DESCRIPTION:
IncobotulinumtoxinA (Xeomin) is a botulinum toxin type A preparation free of complexing proteins. Injected into a muscle, incobotulinumtoxinA causes a reversible local weakening of the muscle for several months, and may improve an impaired muscle function by lessening the muscle tightness within few days. IncobotulinumtoxinA is widely used for various severe neurological conditions. There is some evidence that the treatment effect may be influenced by the amount of the solvent in which incobotulinumtoxinA is diluted before injection.

ELIGIBILITY:
Main Inclusion Criteria:

* Female or male patients ≥ 18 years
* Stable upper limb spasticity of diverse etiology
* Focal spasticity with equal or more than 2 points on the Ashworth scale in the wrist flexors
* Disability Assessment Scale (DAS) ≥ 2 points for primary therapeutic target at both screening and baseline visits

Main Exclusion Criteria:

* Fixed contracture
* Bilateral upper limb paresis/paralysis
* Previous treatment with BoNT of any serotype and for any body region within the 4 months prior to screening
* Previous or planned treatment with phenol- or alcohol-injection in the target limb
* Other muscle hypertonia (e.g. rigidity)
* Diagnosis of myasthenia gravis, Lambert-Eaton-Syndrome, amyotrophic lateral sclerosis, or any other significant neuromuscular disease which might interfere with the study
* Severe atrophy of the target limb muscles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2007-02; Primary Completion 2008-01 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Barnes, MD, FRCP, Principal Investigator — Hunters Moor Hospital, Newcastle-upon-Tyne, UK
Locations (27):
- Austria (3):
  - Hermagor
  - Innsbruck
  - Vienna
- France (4):
  - Besançon
  - Garches
  - Lille
  - Paris
- Germany (3):
  - Beelitz-Heilstätten
  - Düsseldorf
  - Gladbeck
- Italy (6):
  - Bari
  - Costa Masnaga
  - Messina
  - Mestre
  - Milan
  - Rome
- Portugal (2):
  - Lisbon
  - Tocha
- Spain (3):
  - Barcelona
  - Madrid
  - Terrassa
- Switzerland (2):
  - Bern
  - Nottwil
- United Kingdom (4):
  - Kent
  - Liverpool
  - Plymouth
  - Wakefield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 216 female and male subjects with upper limb spasticity caused by either stroke, brain injury, spinal cord injury, multiple sclerosis or cerebral palsy were screened starting February 2007. Recruitment advertisements according to local law and approved by the responsible IEC were published as needed.
Pre-assignment Details: The protocol contained a screening period of 7 days to allow evaluation of laboratory and ECGs in order to determine eligibility. 24 subjects were screening failures due to violation of selection or protocol criteria.
Period: Overall Study
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Started | 97 | 95
Completed | 91 | 89
Not Completed | 6 | 6
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Other | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL | Total
Number analyzed (Participants) | 97 | 95 | 192
Age Continuous [Mean (Standard Deviation); unit: years] | 55.3 (14.88) | 55.5 (13.74) | 55.4 (14.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 33 | 81
  Male | 49 | 62 | 111
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 76 | 78 | 154
  Asian | 0 | 0 | 0
  Oriental | 1 | 0 | 1
  Negroid | 1 | 0 | 1
  Other | 1 | 1 | 2
  Missing | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Responder in Disability Assessment Scale (DAS) at Week 4 - Per Protocol Set
Description: The primary efficacy endpoint is the number of responder at Week 4; response defined as an improvement (reduction) of at least one point in the DAS for the primary therapeutic target from baseline visit to Week 4. The DAS determines the functional impairment for the domains hygiene, dressing, limb position and pain according to the following scale: 0 = no disability; 1 = mild disability; 2 = moderate disability; 3 = severe disability. At Screening visit, the subject and investigator, selected together one of the four domains as the primary therapeutic target.
Time Frame: At week 4
Population: Analysis is based on Per Protocol Set, defined as all randomized subjects who received at least one dose of study drug and who have no major deviation from study protocol. For this set of subjects no missing values can occur for the primary endpoint.
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 81 | 84
participants | 51 | 44
Statistical Analysis 1: Comparison: incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL vs incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL; Null hypothesis: The response rate for the low volume dilution group (50 U/ml) is greater than the response rate for the high volume dilution group (20 U/ml); Test type: Non-Inferiority or Equivalence — A two-sided 95% Newcombe-Wilson confidence interval for the difference between the response rates of the groups was calculated. The lower bound of the Newcombe-Wilson CI for the difference of proportions was compared to the non-inferiority margin of -25%; difference in response rates = 10.6, 95% CI 2-sided [-4.4 to 24.9] — difference in response rates = response rate for high volume dilution group (20 U/ml) - response rate for low volume dilution group (50 U/ml)

2. Secondary Outcome: Responder in DAS at Week 4 - Full Analysis Set
Description: Response is defined as an improvement (reduction) of at least one point in the DAS for the primary therapeutic target from baseline visit.
Time Frame: week 4
Population: Analysis is based on Full Analysis Set, defined as all randomized subjects who received at least one dose of study drug. Missing values were not imputed.
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 94 | 95
participants | 59 | 49

3. Secondary Outcome: Responder in DAS at Week 12 - Full Analysis Set
Description: as for outcome 2
Time Frame: week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 94 | 95
participants | 46 | 38

4. Secondary Outcome: Responder in DAS at Follow up - Full Analysis Set
Description: as for outcome 2
Time Frame: follow up visit, between week 12 and week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 75 | 71
participants | 40 | 33

5. Secondary Outcome: Responder in Frenchay Arm Test (FAT) at Week 4 - Full Analysis Set
Description: Response is defined as an improvement (increase) of at least one point in the FAT from baseline visit. For the FAT the investigator assessed the extent of functionality of the upper limb according to five standardized tests. Each test is rated with 0 = failed or 1 = successfully passed. For the evaluation, the sum of all test scores was calculated resulting in a total score from 0 to 5.
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 94 | 95
participants | 17 | 24

6. Secondary Outcome: Responder in FAT at Week 12 - Full Analysis Set
Description: as for outcome 5
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 94 | 95
participants | 20 | 22

7. Secondary Outcome: Responder in FAT at Follow up - Full Analysis Set
Description: as for outcome 5
Time Frame: follow up visit, between week 12 and week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 75 | 71
participants | 12 | 15

8. Secondary Outcome: Responder in Ashworth Scale (Elbow Flexors) at Week 4 - Full Analysis Set
Description: Response is defined as an improvement of at least one point in the Ashworth Scale for the treated muscle group from baseline visit. The Ashworth Scale is a 5-point-scale to rate to degree of spasticity: 0 = No increase in tone; 1 = Slight increase in tone giving a "catch" when the limb was moved in flexion or extension; 2 = More marked increase in tone, but limb easily flexed; 3 = Considerable increase in tone - passive movements difficult; 4 = Limb rigid in flexion or extension.
Time Frame: week 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 75 | 81
participants | 47 | 50

9. Secondary Outcome: Responder in Ashworth Scale (Elbow Flexors) at Week 12 - Full Analysis Set
Description: Response is defined as an improvement of at least one point in the Ashworth Scale for the treated muscle group from baseline visit.
Time Frame: week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 75 | 81
participants | 37 | 40

10. Secondary Outcome: Responder in Ashworth Scale (Elbow Flexors) at Follow up - Full Analysis Set
Description: as for outcome 9
Time Frame: follow up visit, between week 12 and week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 59 | 62
participants | 30 | 21

11. Secondary Outcome: Responder in Ashworth Scale (Wrist Flexors) at Week 4 - Full Analysis Set
Description: as for outcome 9
Time Frame: week 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 87 | 89
participants | 68 | 63

12. Secondary Outcome: Responder in Ashworth Scale (Wrist Flexors) at Week 12 - Full Analysis Set
Description: as for outcome 9
Time Frame: week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 87 | 89
participants | 43 | 46

13. Secondary Outcome: Responder in Ashworth Scale (Wrist Flexors) at Follow up - Full Analysis Set
Description: as for outcome 9
Time Frame: follow up visit, between week 12 and week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 69 | 67
participants | 31 | 28

14. Secondary Outcome: Responder in Ashworth Scale (Thumb Flexors) at Week 4 - Full Analysis Set
Description: as for outcome 9
Time Frame: week 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 35 | 32
participants | 29 | 19

15. Secondary Outcome: Responder in Ashworth Scale (Thumb Flexors) at Week 12 - Full Analysis Set
Description: as for outcome 9
Time Frame: week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 35 | 32
participants | 21 | 13

16. Secondary Outcome: Responder in Ashworth Scale (Thumb Flexors) at Follow up - Full Analysis Set
Description: as for outcome 9
Time Frame: follow up visit, between week 12 and week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 30 | 23
participants | 18 | 9

17. Secondary Outcome: Responder in Ashworth Scale (Fingers Flexors) at Week 4 - Full Analysis Set
Description: as for outcome 9
Time Frame: week 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 78 | 81
participants | 57 | 48

18. Secondary Outcome: Responder in Ashworth Scale (Fingers Flexors) at Week 12 - Full Analysis Set
Description: as for outcome 9
Time Frame: week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 78 | 81
participants | 35 | 35

19. Secondary Outcome: Responder in Ashworth Scale (Fingers Flexors) at Follow up - Full Analysis Set
Description: as for outcome 9
Time Frame: follow up visit, between week 12 and week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 62 | 60
participants | 17 | 20

20. Secondary Outcome: Responder in Ashworth Scale (Forearm Pronators) at Week 4 - Full Analysis Set
Description: as for outcome 9
Time Frame: week 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 42 | 46
participants | 32 | 30

21. Secondary Outcome: Responder in Ashworth Scale (Forearm Pronators) at Week 12 - Full Analysis Set
Description: as for outcome 9
Time Frame: week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 42 | 46
participants | 28 | 22

22. Secondary Outcome: Responder in Ashworth Scale (Forearm Pronators) at Follow up - Full Analysis Set
Description: as for outcome 9
Time Frame: follow up visit, between week 12 and week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 34 | 36
participants | 18 | 16

23. Secondary Outcome: Change From Baseline in Passive Range of Motion (PROM) - Wrist Extension
Description: For the PROM all motions of wrist and elbow were measured from a defined neutral starting point position. The degrees of motion were added in the direction the wrist and elbow moved from the neutral starting position. The neutral starting position was the position of an upright standing/sitting person. The angle of the motion from the neutral starting position was measured in degrees using a goniometer. Angles were measured for the wrist with maximal dorsal extension, neutral position and maximal palmar flexion, and for the elbow with maximal extension, neutral position and maximal flexion.
Time Frame: baseline, week 4, week 12, follow up (between week 12 and week 20)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: degree
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 97 | 95
degree
  Week 4 | 14.8 (3.31) [-10.3 to 8.7] | 15.7 (3.47) [-10.3 to 8.7]
  Week 12 | 7.3 (3.15) [-12.2 to 5.9] | 10.4 (3.32) [-12.2 to 5.9]
  Follow up (between week 12 and week 20) | 8.2 (4.62) [-15.6 to 11.2] | 10.4 (4.93) [-15.6 to 11.2]

24. Secondary Outcome: Change From Baseline in Passive Range of Motion (PROM) - Elbow Extension
Description: as for outcome 23
Time Frame: baseline, week 4, week 12, follow up (between week 12 and week 20)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: degree
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 97 | 95
degree
  Week 4 | 8.0 (3.37) [-7.3 to 11.7] | 5.8 (3.42) [-7.3 to 11.7]
  Week 12 | 6.1 (4.50) [-8.5 to 16.6] | 2.1 (4.46) [-8.5 to 16.6]
  Follow up (between week 12 and week 20) | 3.9 (3.58) [-10.3 to 9.8] | 4.1 (3.58) [-10.3 to 9.8]

25. Secondary Outcome: Change From Baseline in Passive Range of Motion (PROM) - Wrist Maximum Flexion
Description: as for outcome 23
Time Frame: baseline, week 4, week 12, follow up (between week 12 and week 20)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: degree
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 97 | 95
degree
  Week 4 | -1.2 (2.34) [-13.1 to 0.3] | 5.2 (2.45) [-13.1 to 0.3]
  Week 12 | -1.3 (2.48) [-11.3 to 3.0] | 2.9 (2.62) [-11.3 to 3.0]
  Follow up (between week 12 and week 20) | -1.3 (2.62) [-12.7 to 2.5] | 3.8 (2.80) [-12.7 to 2.5]

26. Secondary Outcome: Change From Baseline in Passive Range of Motion (PROM) - Elbow Maximum Flexion
Description: as for outcome 23
Time Frame: baseline, week 4, week 12, follow up (between week 12 and week 20)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: degree
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 97 | 95
degree
  Week 4 | 0.1 (2.60) [-9.9 to 4.6] | 2.7 (2.60) [-9.9 to 4.6]
  Week 12 | -0.7 (2.45) [-10.1 to 3.5] | 2.6 (2.41) [-10.1 to 3.5]
  Follow up (between week 12 and week 20) | -1.9 (2.86) [-10.8 to 5.1] | 1.0 (2.81) [-10.8 to 5.1]

27. Secondary Outcome: Investigator's Global Assessment of Treatment Response (GATR) - Full Analysis Set
Description: The investigator's global assessment of response to treatment were determined with the use of the Global Response Scale using the following scores: -4 = very marked worsening; -3 = marked worsening; -2 = moderate worsening; -1 = mild worsening; 0 = no change; +1 = mild improvement; +2 = moderate improvement; +3 = marked improvement; +4 = very marked improvement.
Time Frame: week 4
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 97 | 95
units on a scale | 1.66 (0.106) | 1.59 (0.106)

28. Secondary Outcome: Patient's Global Assessment of Treatment Response (GATR) - Full Analysis Set
Description: The patient's global assessment of response to treatment were determined with the use of the Global Response Scale using the following scores: -4 = very marked worsening; -3 = marked worsening; -2 = moderate worsening; -1 = mild worsening; 0 = no change; +1 = mild improvement; +2 = moderate improvement; +3 = marked improvement; +4 = very marked improvement.
Time Frame: week 4
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 97 | 95
units on a scale | 1.41 (0.121) | 1.48 (0.121)

29. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Week 4 - Item Feeding
Description: Response is defined as an improvement (increase) of at least one point in the Barthel Index from baseline visit. The Barthel Index was assessed for the items feeding, grooming, toilet use, bathing and dressing. Feeding: 0 = unable; 1 = needs help cutting, spreading butter etc.; 2 = independent; Grooming: 0 = needs help with personal care; 1 = independent face/hair/teeth/shaving; Toilet use: 1 = need some help, but could do something alone; 2 = independent; Bathing: 0 = dependent; 1 = independent; Dressing: 0 = dependent; 1 = needs help but could do about half unaided; 2 = independent.
Time Frame: week 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 94 | 95
participants | 7 | 5

30. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Week 12 - Item Feeding
Description: as for outcome 29
Time Frame: week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 94 | 95
participants | 8 | 6

31. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Follow up - Item Feeding
Description: as for outcome 29
Time Frame: follow up visit, between week 12 and week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 75 | 71
participants | 7 | 5

32. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Week 4 - Item Grooming
Description: as for outcome 29
Time Frame: week 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 94 | 95
participants | 5 | 6

33. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Week 12 - Item Grooming
Description: as for outcome 29
Time Frame: week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 94 | 95
participants | 7 | 10

34. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Follow up - Item Grooming
Description: as for outcome 29
Time Frame: follow up visit, between week 12 and week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 75 | 71
participants | 7 | 6

35. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Week 4 - Item Toilet Use
Description: as for outcome 29
Time Frame: week 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 94 | 95
participants | 7 | 6

36. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Week 12 - Item Toilet Use
Description: as for outcome 29
Time Frame: week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 94 | 95
participants | 11 | 7

37. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Follow up - Item Toilet Use
Description: as for outcome 29
Time Frame: follow up visit, between week 12 and week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 75 | 71
participants | 11 | 5

38. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Week 4 - Item Bathing/Showering
Description: as for outcome 29
Time Frame: week 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 94 | 95
participants | 1 | 7

39. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Week 12 - Item Bathing/Showering
Description: as for outcome 29
Time Frame: week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 94 | 95
participants | 4 | 6

40. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Follow up - Item Bathing/Showering
Description: as for outcome 29
Time Frame: follow up visit, between week 12 and week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 75 | 71
participants | 2 | 4

41. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Week 4 - Item Dressing
Description: as for outcome 29
Time Frame: week 4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 94 | 95
participants | 9 | 6

42. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Week 12 - Item Dressing
Description: as for outcome 29
Time Frame: week 12
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 94 | 95
participants | 10 | 8

43. Secondary Outcome: Response Rates in Activity of Daily Living (Barthel Index) at Follow up - Item Dressing
Description: as for outcome 29
Time Frame: follow up visit, between week 12 and week 20
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Number analyzed (Participants) | 75 | 71
participants | 8 | 7

ADVERSE EVENTS:
Time Frame: All SAEs/AEs up to 20 weeks after injection
Description: The investigator asked the patient for AEs systematically at each visit.
  The table of "Other Adverse Events" includes all non-serious AEs.
  The Safety Analysis Set differs from the Full Analysis Set due to a randomization error (one patient randomized to low dilution in fact received high dilution).
Arm/Group | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL
Serious Adverse Events (participants affected / at risk) | 6/96 | 6/96
Other Adverse Events (participants affected / at risk) | 15/96 | 17/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL (N=96) | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL (N=96)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cerebral hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0)
Epileptic Aura (Nervous system disorders) | 0 (0) | 1 (2)
Fecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) — abdominal pain due to concomitant coprostasis
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Visual disturbance (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | incobotulinumtoxinA (Xeomin) High-volume Dilution 20 Units/mL (N=96) | incobotulinumtoxinA (Xeomin) Low-volume Dilution 50 Units/mL (N=96)
Bronchitis (Infections and infestations) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Epilepsy (Nervous system disorders) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Headache (Nervous system disorders) | 2 | 0
Haematoma (Vascular disorders) | 0 | 2
Injection site haematoma (General disorders) | 0 | 4
Injection site pain (General disorders) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 4
Pain (General disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No results to be published without written agreement by sponsor; manuscripts to be sent to sponsor at least 6 weeks before submission. Sponsor to give written opinion within 30 days. Sponsor is entitled to exert influence on the contents of publications, to postpone publications up to 36 months after end of the study, and to name co-authors. In case of justified doubts of sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.